CLINICAL TRIAL: NCT03991754
Title: Usefulness of Amiodarone for the Prevention of New Onset Atrial Fibrillation After Transcatheter Aortic Valve Implantation: a Randomized Controlled Trial
Brief Title: Prevention of New Onset AF After TAVI (PAF-TAVI Trial)
Acronym: PAF-TAVI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luis Nombela Franco (Other)
Responsible Party: Sponsor-Investigator, Luis Nombela Franco, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19/147-R_M
Record Dates: First submitted 2019-05-30; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation New Onset
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Phase III Clinical trial, multiple sites, controlled, randomized, double blind, parallel groups.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiodarone (Experimental): Oral Amiodarone 600mg / day, divided into 3 doses (200mg every 8 hours) for 6 days before the procedure and then 400mg / day, divided into 2 doses (200mg every 12 hours) during the 6 days following the implantation of TAVI.
  Interventions: Procedure: transcatheter aortic valve implantation
- Control (Placebo Comparator): Patients assigned to the control group will receive placebo tablets identical to those of amiodarone. The administration of these tablets will follow the same scheme as in the amiodarone group. Therefore, they will receive placebo tablets orally, 1 tablet every 8 hours 6 days before the procedure and then 1 tablet every 12 hours during the 6 days following the implantation of TAVI
  Interventions: Procedure: transcatheter aortic valve implantation

INTERVENTIONS:
Procedure: transcatheter aortic valve implantation — transcatheter aortic valve implantation

SUMMARY:
New onset atrial fibrillation (NOAF) is a relatively frequent complication after transcatheter aortic valve implantation (TAVI). This complication has been related with worse short and long-term outcomes, including higher stroke, mortality, readmission and bleeding rates. The aim of this study is to evaluate the effectiveness of amiodarone in the prevention of the NOAF after TAVI.

The study is a multicenter, randomized double-blinded trial including 120 patients without prior AF that will undergo TAVI in a scheduled basis. Patients will be randomized to be treated with amiodarone orally from 6 days before to 6 days after the TAVI procedure versus placebo.

All the patients will be monitored with a 60-day holter to evaluate NOAF incidence. The main objective is NOAF incidence after TAVI at 30-day. Secondary endpoints are the incidence of NOAF, stroke, bleeding and all-cause and cardiovascular mortality in both groups at 60-day. Results of this study can contribute to optimize TAVI results in a short and long term, potentially improving the survival and quality of life in this group of frail patients with comorbidities, which makes them vulnerable to NOAF, stroke, bleeding, heart failure and readmission.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old. Women of childbearing age must commit to the use of contraceptive methods of assured efficacy.
* Patients that will undergo TAVI due to aortic stenosis.
* Sinus rhythm showed by an ECG during 72 hours previous to the inclusion in the study.

Exclusion Criteria:

* Pregnancy or lactation. Women of childbearing age who do not have a negative pregnancy test.
* Paroxysmal persistent or persistent AF (documented record in electrocardiogram or ECG holter)
* Congestive heart failure with functional class NYHA IV despite optimal medical treatment.
* Sustained hypotension (TAS < 80mmHg)
* Severe mitral stenosis or regurgitation
* Treatment with antiarrhythmic drugs (amiodarone included) 3 months before the procedure, treatment with beta-blockers or dihydropyrimidine calcium channel blockers are not considered an exclusion criteria.
* Sinus bradycardia (< 50 lpm), PR interval >240 mseg or second or third degree AV block.
* QT interval longer than 480 msec in an EKG performed in 72 hours before the inclusion, without a permanent pacemaker.
* Clinical hypo- or hyperthyroidism, clinical or subclinical autoimmune thyroid disease, or multinodular goiter.
* Allergy or adverse reaction known or suspected to the amiodarone.
* Denial of the patient or inability to give informed consent.
* Hypersensitivity to iodo
* Concomitant drugs that, in association with amiodarone, can induce torsades de pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of new onset atrial fibrillation | 30 days after transcatheter aortic valve implantation (TAVI)
  Compare the incidence of new onset atrial fibrillation (NOAF) on patients that receive oral amiodarone versus placebo. NOAF is defined as an irregular rhythm without P wave and irregular ventricular response during at least 30 seconds, detected in the electrocardiographic monitoring during the post-procedural period or in the 60 days ECG Holter in a patient without previous history of atrial fibrillation. NOAF incidence within 30-day after the TAVI procedure is the primary end-point.

SECONDARY OUTCOMES:
Incidence of new onset atrial fibrillation | 60 days after transcatheter aortic valve implantation (TAVI)
  Compare the incidence of new onset atrial fibrillation (NOAF) on patients that receive oral amiodarone versus placebo. NOAF is defined as an irregular rhythm without P wave and irregular ventricular response during at least 30 seconds, detected in the electrocardiographic monitoring during the post-procedural period or in the 60 days ECG Holter in a patient without previous history of atrial fibrillation. NOAF incidence within 30-day after the TAVI procedure is the primary end-point.
Effect of the amiodarone | 1-year follow-up
  Analyze the effect of the amiodarone in the moment of appearance and the burden of AF after TAVI. AF burden, defined as the relative length of the AF registers in relation to the time in sinus rhythm.
Mortality and CV mortality. | 1-year follow-up
  Compare all-cause mortality and CV mortality between groups.
Number of parients with MACE | at 30 days after NOAF
  MACE: Stroke, bleeding (major or life-threatening), and all-cause and cardiovascular mortality rate.
Number of parients with MACE | at 60 days after NOAF
  MACE: Stroke, bleeding (major or life-threatening), and all-cause and cardiovascular mortality rate.
Number of parients with MACE | at 6 months after NOAF
  MACE: Stroke, bleeding (major or life-threatening), and all-cause and cardiovascular mortality rate.
Number of parients with MACE | 1-year follow-up
  MACE: Stroke, bleeding (major or life-threatening), and all-cause and cardiovascular mortality rate.
Number of adverse events related to amiodarone | at 30 days after NOAF
  The safety evaluation will be realized by a meticulous vigilance of the adverse effects appeared in the study population.
Number of adverse events related to amiodarone | at 60 days after NOAF
  The safety evaluation will be realized by a meticulous vigilance of the adverse effects appeared in the study population.
Number of adverse events related to amiodarone | at 6 months after NOAF
  The safety evaluation will be realized by a meticulous vigilance of the adverse effects appeared in the study population.
Number of adverse events related to amiodarone | 1-year follow-up
  The safety evaluation will be realized by a meticulous vigilance of the adverse effects appeared in the study population.
Incidence of permanent pacemaker implantation in the both groups. | at 30 days after NOAF
  Need of permanent pacemaker implantation in the both groups.
Incidence of permanent pacemaker implantation in the both groups. | at 60 days after NOAF
  Need of permanent pacemaker implantation in the both groups.
Incidence of permanent pacemaker implantation in the both groups. | at 6 months after NOAF
  Need of permanent pacemaker implantation in the both groups.
Incidence of permanent pacemaker implantation in the both groups. | 1-year follow-up
  Need of permanent pacemaker implantation in the both groups.
Quality of life: EuroQoL 5D | at 30 days after NOA
  Eq-5D: EuroQoL 5 Dimensions. Score between 0 and 1. The best score 1.
Quality of life: Kansas City test | at 30 days after NOA
  Score between 0 and 100. The best score 100.
Quality of life: EuroQoL 5D | at 60 days after NOAF
  Eq-5D: EuroQoL 5 Dimensions. Score between 0 and 1. The best score 1.
Quality of life: Kansas City test | at 60 days after NOAF
  Score between 0 and 100. The best score 100.
Quality of life: EuroQoL 5D | at 6 months after NOAF
  Eq-5D: EuroQoL 5 Dimensions. Score between 0 and 1. The best score 1.
Quality of life: Kansas City test | at 6 months after NOAF
  Score between 0 and 100. The best score 100.
Quality of life: EuroQoL 5D | 1-year follow-up
  Eq-5D: EuroQoL 5 Dimensions. Score between 0 and 1. The best score 1.
Quality of life: Kansas City test | 1-year follow-up
  Score between 0 and 100. The best score 100.
Readmissions due to CV causes | 1-year follow-up
  Compare the number of readmissions due to CV causes
Functional change: New York Heart Association. | at 30 days after NOA
  Evaluate the functional change according to the NYHA scale. Score between 0 and 4. The best score 1.
Functional change: New York Heart Association. | at 60 days after NOAF
  Evaluate the functional change according to the NYHA scale. Score between 0 and 4. The best score 1.
Functional change: New York Heart Association. | at 6 months after NOAF
  Evaluate the functional change according to the NYHA scale. Score between 0 and 4. The best score 1.
Functional change: New York Heart Association. | 1-year follow-up
  Evaluate the functional change according to the NYHA scale. Score between 0 and 4. The best score 1.
Capacity for the exercise | at 30 days after NOA
  Evalue the change in capacity for the exercise, evaluated by the 6-minute walk test between groups
Capacity for the exercise | at 60 days after NOAF
  Evalue the change in capacity for the exercise, evaluated by the 6-minute walk test between groups
Capacity for the exercise | at 6 months after NOAF
  Evalue the change in capacity for the exercise, evaluated by the 6-minute walk test between groups
Capacity for the exercise | 1-year follow-up
  Evalue the change in capacity for the exercise, evaluated by the 6-minute walk test between groups
Incidence of Acute renal failure | baseline
  Compare the number of events due to acute renal failure between groups
Incidence of Acute renal failure | 30 days after NOA
  Compare the number of events due to acute renal failure between groups